CLINICAL TRIAL: NCT02800590
Title: A Phase II, Two-part, Multiple-dose, Dose-finding, Single-blind Study to Investigate the Safety and Efficacy of ABP-700 for Procedural Sedation in Adult Patients Undergoing Colonoscopy
Brief Title: Study to Investigate the Safety and Efficacy of 3 Dosing Regimens of ABP-700 for Procedural Sedation in Adult Participants Undergoing Colonoscopy
Acronym: ABP-700
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MDCO-ABP-15-01; 2015-004019-19 (EudraCT Number)
Record Dates: First submitted 2016-06-10; First posted 2016-06-15 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Colonoscopy
Keywords: Adult participants; Sedation; elective
MeSH Terms: interventions — abp-700

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABP-700 30 μg/kg/min (Experimental): Starting intravenous (IV) infusion rate of 50 micrograms per kilogram per minute (μg/kg/min) for 5 minutes, followed by 30 μg/kg/min until the procedure is complete. Up to 2 supplemental bolus injections of 50 μg/kg ABP-700 separated by a minimum of 5 minutes may be administered in order to achieve and/or maintain adequate procedure conditions.
  Interventions: Drug: ABP-700
- ABP-700 40 μg/kg/min (Experimental): Starting IV infusion rate of 70 μg/kg/min for 3 minutes, followed by 40 μg/kg/min until the procedure is complete. Up to 2 supplemental bolus injections of 50 μg/kg ABP-700 separated by a minimum of 5 minutes may be administered in order to achieve and/or maintain adequate procedure conditions.
  Interventions: Drug: ABP-700
- ABP-700 45 μg/kg/min (Experimental): Starting IV infusion rate of 80 μg/kg/min for 3 minutes, followed by 45 μg/kg/min until the procedure is complete. Up to 2 supplemental bolus injections of 50 μg/kg ABP-700 separated by a minimum of 5 minutes may be administered in order to achieve and/or maintain adequate procedure conditions.
  Interventions: Drug: ABP-700

INTERVENTIONS:
Drug: ABP-700

SUMMARY:
This is a phase II, two-part, multiple-dose, dose-finding, single-blind study in adult participants undergoing elective colonoscopy for screening or diagnostic purposes. This study is designed to test various ABP-700 infusion regimens for rational selection of one or more dosage regimen(s) to be used for future clinical development of ABP-700 in procedural sedation.

DETAILED DESCRIPTION:
In Part 1, three ABP-700 two-stage infusion regimens will be evaluated. A sample size of 75 evaluable participants will be randomly assigned to dose regimens in a 1:1:1 ratio. Following the completion of Part 1, a Data Review Committee (DRC) will review the dose-response, efficacy, and safety data and provide recommendations on whether to continue the study to Part 2 and the number of ABP-700 infusion regimens to be included in Part 2. The Sponsor (MDCO) will make the final decision to proceed with Part 2 (whether to conduct Part 2 and number of dose regimens if the study continues to Part 2) based on the recommendation from the DRC.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be male or female 18 to 75 years of age, inclusive
* Participant must give written informed consent before initiation of any study-related procedures
* Participant is scheduled to undergo elective colonoscopy
* Body Mass Index (BMI) 18.0 to 29.0 kilogram per meter squared (kg/m^2)
* American Society of Anesthesiology (ASA) class I to II
* Modified Mallampati score I to II
* If female and of child-bearing potential, participant must have a negative pregnancy test during screening and cannot be breast-feeding
* If participant is a sexually active male or a sexually active female of child-bearing potential, he or she must agree to use a medically accepted form of contraception from the time of consent to completion of all follow-up study visits

Exclusion Criteria:

* Any ASA physical status III or worse, or history of one or more of the following: history or presence of significant cardiovascular disease, including atrial fibrillation or cardiovascular disease risk factors, hyperlipidemia, coronary artery disease, or any known genetic pre disposition to cardiac arrhythmia (including long QT syndrome, > 450 milliseconds [msec]); history of any neurological or seizure disorder or psychiatric disease; history or presence of significant pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic or dermatologic disease; history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the participant by their participation in the study.
* History of any recent illness (such as, upper respiratory infection) that does not satisfy ASA III or greater requirements but in the opinion of the investigator, may pose an additional risk to the participant by their participation in the study.
* Participants with a history of essential hypertension that are not well controlled on medication will be accepted. Participants should have been diagnosed with hypertension for at least 6 months and/or are not on stable therapy for at least 4 weeks prior to the study.
* Surgery within the past 90 days prior to dosing judged by the investigator to be clinically relevant.
* History of febrile illness within 5 days prior to dosing.
* Participants in whom airway management is judged to be potentially difficult; thyromental distance ≤ 4 centimeters (cm) or Mallampati scores of 3 or 4 or per the discretion of the anesthesiologist based on history and physical exam.
* History or presence of alcoholism, drug abuse, or illicit drug use within the past 2 years.
* Hypersensitivity or idiosyncratic reaction to components of ABP-700 (sulfobutylether-beta-cyclodextrin, citrate buffer, sodium hydroxide), remifentanil or midazolam.
* Participant is the investigator or his/her deputy, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the study.
* Participation in another interventional clinical trial within 90 days prior to dosing. The 90-day window will be derived from the date of the last study procedure (such as last blood collection or dosing) in the previous study to Day 1 of the current study.
* Participants who, for any reason, are deemed by the investigator to be inappropriate for this study, including participants who are unable to communicate or to cooperate with the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of Successfully Completed Procedures by Assigned ABP-700 Infusion Dose | Treatment period (Day 1)

SECONDARY OUTCOMES:
Number of Successfully Completed Procedures by Assigned ABP-700 Infusion Dose with and without Supplemental Bolus ABP-700 | Treatment period (Day 1)
Number of Successfully Completed Procedures by Assigned ABP-700 Infusion Dose with and without Supplemental Bolus ABP-700 that Require or Do Not Require Rescue Sedative Medication | Treatment period (Day 1)
Time to Procedure Start | Treatment period (Day 1)
Depth and Duration of Sedation | Treatment period (Day 1)
Number of Supplemental ABP-700 Bolus Doses Required | Treatment period (Day 1)
Recovery from Sedation and Discharge Conditions as Assessed by the Modified Aldrete Score (APRS) | Treatment period (Day 1)

CONTACTS AND LOCATIONS:
Overall Officials: A.R. Absalom, MD, Principal Investigator — University Medical Center Groningen (UMCG)
Locations (3):
- Netherlands (3):
  - Martini Hospital, Groningen
  - University Medical Center Groningen (UMCG), Groningen
  - Radboud University Nijmegen Medical Centre, Nijmegen

IPD SHARING:
Plan to Share IPD: No